CLINICAL TRIAL: NCT06880419
Title: A Prospective, Single-arm, Historically Controlled, Single-center Study for Preventing aGVHD, Post-allogeneic HSCT, in Adults at Moderate-to-high Risk Using Recombinant Humanized Anti-CD25 Monoclonal Antibody Based on the daGOAT Model
Brief Title: Anti-CD25 rhMAb for aGVHD Prevention in High-Risk Adults Using the daGOAT Model
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT2024115
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Acute Graft-versus-Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group of daGOAT model prevention (Experimental): Model-predicted patients at high risk (HR): Recombinant humanized anti-CD25 monoclonal antibody: 50 mg/day when the post-transplant model predicts high risk in the second week post-prediction and 25 mg/day in the fourth and sixth weeks post-prediction. Administered in combination with conventional aGVHD prevention regimen.
  Model-predicted patients at moderate risk (MR): Recombinant anti-CD25 humanized monoclonal antibody: 25 mg/day when the model predicts intermediate risk post-transplantation and at the 2nd, 4th, and 6th weeks post-prediction. Administered in combination with conventional aGVHD prevention regimen.
  Model-predicted patients at low-risk (LR): A conventional aGVHD prevention regimen only was used.
  Interventions: Drug: Recombinant Humanized Anti-CD25 Monoclonal Antibody Injection

INTERVENTIONS:
Drug: Recombinant Humanized Anti-CD25 Monoclonal Antibody Injection — Model-predicted patients at high risk (HR): Recombinant humanized anti-CD25 monoclonal antibody: 50 mg/day when the post-transplant model predicts high risk in the second week post-prediction and 25 mg/day in the fourth and sixth weeks post-prediction. Administered in combination with conventional aGVHD prevention regimen.
  Model-predicted patients at moderate risk (MR): Recombinant anti-CD25 humanized monoclonal antibody: 25 mg/day when the model predicts intermediate risk post-transplantation and at the 2nd, 4th, and 6th weeks post-prediction. Administered in combination with conventional aGVHD prevention regimen.
  Model-predicted patients at low-risk (LR): A conventional aGVHD prevention regimen only was used.

SUMMARY:
To assess the efficacy and safety of using recombinant humanized anti-CD25 monoclonal antibody injection as a prophylactic strategy for reducing the incidence of severe acute graft-versus-host disease (aGVHD) in adult patients at intermediate to high risk, as predicted by the dynamic aGVHD Onset Anticipation Tianjin (daGOAT) model, following allogeneic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years, regardless of gender.
2. Patients with hematologic disorders who are scheduled to receive allo-HSCT.
3. Voluntarily join this study, sign the informed consent form, have good compliance, and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients who have received a second or multiple transplants.
2. Patients who are allergic to, or intolerant of, a recombinant humanized anti-CD25 monoclonal antibody injection.
3. Pregnant or lactating female patients or female patients who are unable to take effective contraceptive measures during the entire trial period.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe aGVHD (Grade III-IV) within 100 days post-transplantation | 100 days after transplantation

SECONDARY OUTCOMES:
Incidence of aGVHD and aGVHD (any grade) in each target organ within 100 days post-transplantation | 100 days after transplantation
Engraftment rate | 180 days after transplantation
Disease relapse rate | 180 days after transplantation
Infection rate | 180 days after transplantation
Overall survival | 180 days after transplantation
Non-relapse mortality | 180 days after transplantation
GVHD-free relapse-free survival | 180 days after transplantation
Overall Response Rate of severe aGVHD treatment | 100 days after transplantation
Incidence of chronic GVHD | 180 days after transplantation
Adverse events | 180 days after transplantation
Total cost of treatment | 180 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No